CLINICAL TRIAL: NCT03119922
Title: National Project for Healthcare Assessment of SCD Children Diagnosed by Newborn Screening in France
Brief Title: Quality of Care of Children With Sickle Cell Disease (SCD) Screened at Birth in France
Acronym: EVADREP
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: CNAMTS (Unknown); AFDPHE (Unknown); National reference center for thalassemia (Unknown); National laboratories in charge of the SCD new born screening (Unknown); Reference and competence centers for RBC disorders (Unknown)
Responsible Party: Sponsor
Other Study IDs: NI 12001
Record Dates: First submitted 2017-01-10; First posted 2017-04-19 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2016-12

CONDITIONS: New-borns Screening; Sickle Cell Disease
Keywords: major sickle cell disease (SCD); children; pneumococcal preventive measures
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SCD french new born: New-borns diagnosed by NBS from 01/01/2006 to 31/12/2010 (AFDPHE data, France)
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention

SUMMARY:
The main objective of this study is to evaluate at the national level (France)

* the early healthcare practices for children with sickle cell disease screened at birth,
* the adequacy of theses practices with the national recommendations,
* their variability over time and according the characteristics of treatment centers.

Will be studied in particular the diffusion of the latest preventive measures (practice of trans-cranial Doppler and pneumococcal conjugate vaccine) and their link with the residual risks of death, stroke and invasive pneumococcal infections. The study includes all patients born in France between 01/01/2006 and 31/12/2010. Events are recorded and analysed only during the first 5 years of life.

DETAILED DESCRIPTION:
In agreement with the National Insurance Fund (CNAMTS) and the French Association for Screening and Prevention of Child Handicaps (AFDPHE), the French SCD newborn screening (NBS) program is not universal but "targeted" to children identified "at risk" because of the geographical origin of their parents (from a country where the prevalence of sickle cell trait is high: Sub-Saharan Africa, the Caribbean, North Africa, Mediterranean Basin). The number of children diagnosed at birth is increasing steadily each year and sickle cell disease is now in France the most common disease found among those screened in the neonatal period. The total number of new-borns diagnosed by NBS from 01/01/2006 to 31/12/2010 is 1800 (AFDPHE data).

In the absence of preventive care, a high mortality rate is observed during the first 5 years of life, the two main causes of death being invasive pneumococcal infection and splenic sequestration acute. Early care allows to largely preventing invasive pneumococcal disease (by combination of PeniV long-term treatment and pneumococcal vaccinations) and severe acute splenic sequestrations (by establishing a parent education program). Also, prevention of cerebral vascular disease, the most serious complications of sickle cell disease in young children, has been made possible the last 10-15 years by the systematic use of trans-cranial Doppler (TCD). In rich countries, the mortality rate of SCD children detected at birth, is now reduced to less than1-2%. The last French report analysed the results of national NBS program for the period 1995- 2000. Consequently these results did not take into account the most recent advances (use of pneumococcal conjugate vaccine and diffusion of TCD). It is now well demonstrated that these two preventive actions have further improved the morbidity and mortality of children with sickle cell disease.

Recently the French paediatric team from Creteil (France), reported the results of 217 children screened at birth between 1988 and 2007: this single-center study finds excellent results with a 1.9% probability of occurrence of stroke at the age of 18 years for SS and S-Beta0 children. These results should be compared with those obtained for the whole concerned population in France. In order to describe and analyse recent national results on residual morbidity and mortality, the investigators conducted this national retrospective study (EVADREP) studying clinical care during the 5 first years of life of SCD patients diagnosed at birth for the period 2006- 2010.

ELIGIBILITY:
Inclusion Criteria:

* Children born in France (metropolitan France and DOM/TOM) between 01/01/2006 and 31/12/2010
* Identified with a major sickle cell syndrome through national newborn screening .
* All types of major sickle cell disease are concerned: SS, S-Beta0 or +, SC, other (S-O-Arab, S-D Punjab)

Exclusion Criteria:

* Refusal to participate in the study expressed by the holders of parental authority

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: The project is national and aims exhaustiveness of participation of all children diagnosed with major sickle cell syndrome through newborn screening in the period of interest. The choice 2006 - 2010 is justified by the fact that during this recent period, new prevention tools (TCD, Prevenar) were fully available. The upper limit set on 31/12/2010 led for all children to a minimum follow of 3 years,
Sampling Method: Non-Probability Sample
Enrollment: 1750 (Actual)
Dates: Start 2014-03; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Survival at 3 years of age | between 1/01/2014 and 31/12/2015
Probability of survival at 5 years of age | between 1/01/2014 and 31/12/2015
Causes of death | between 1/01/2014 and 31/12/2015

SECONDARY OUTCOMES:
Use of pneumococcal preventive measures: proportion of children who received a full pneumococcal vaccine program (4Prevenar + 1 P23) at 3 and 5 years of age | between 1/01/2014 and 31/12/2015
National diffusion of Trans-cranial Doppler (TCD) : proportion of children who underwent a least one TCD at the age of 2 years and the proportion of children annually monitored | between 1/01/2014 and 31/12/2015
Proportion of children lost to follow-up at birth, at 3 and 5 years of age and reasons for the lack of monitoring | between 1/01/2014 and 31/12/2015
Poportion of patient with current residual risk of stroke and invasive bacterial infections especially pneumococcal infection at 3 years of age | between 1/01/2014 and 31/12/2015
Number of patient with current residual risk of stroke and invasive bacterial infections especially pneumococcal infection at 5 years of age (probability) | between 1/01/2014 and 31/12/2015